CLINICAL TRIAL: NCT06284915
Title: A Parallel-group, Prevention, Phase III, Modified Double-blind, 2-arm, Study to Investigate the Immunogenicity and Describe the Safety of a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW Conjugate Vaccine) Compared With Nimenrix® When Administered in a 1+1 Schedule in Healthy Infants and Toddlers at 6 and 12 Months of Age
Brief Title: Study on Immunogenicity and Safety of a Meningococcal ACYW Conjugate Vaccine in Healthy Infants and Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MEQ00089; 2023-508177-85 (Registry Identifier: CTIS); U1111-1280-6981 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Meningococcal Immunisation; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be performed in a modified double-blind fashion:
  * Investigators and study staff who conduct the safety assessment, and the participants parent/ legally acceptable representative will not know which study intervention is administered
  * Only the study staff who prepare and administer the study intervention and are not involved with the safety evaluation will know which study intervention is administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: MenACYW conjugate vaccine (Experimental): Participants will receive MenACYW Conjugate Vaccine (MenQuadfi®): 2-dose schedule (1+1); dose 1 (priming dose) at 6-7 months of age and dose 2 (booster dose) at 12-13 months of age (MenQuadfi®)
  Interventions: Biological: MenACYW conjugate vaccine
- Group 2: Nimenrix® (Active Comparator): Participants will receive Nimenrix®: 2-dose schedule (1+1); dose 1 (priming dose) at 6-7 months of age and dose 2 (booster dose) at 12-13 months of age
  Interventions: Biological: MenACYW conjugate vaccine

INTERVENTIONS:
Biological: MenACYW conjugate vaccine — Pharmaceutical form:Solution for injection (in a single-dose vial)-Route of administration:Intramuscular (IM) injection
  Other Names: MenQuadfi®
  Arms: Group 1: MenACYW conjugate vaccine
Biological: MenACYW conjugate vaccine — Pharmaceutical form:Solution for injection (powder or cake in a single dose glass vial and a clear and colourless solvent in a pre filled syringe for reconstitution-Route of administration:Intramuscular (IM) injection
  Other Names: Nimenrix®
  Arms: Group 2: Nimenrix®

SUMMARY:
This study is conducted to support a 2-dose series (1+1 vaccination schedule) for immunization of individuals from 6 months of age. The study is designed to evaluate the non-inferiority of the immunological response of MenACYW conjugate vaccine to Nimenrix® after the completion of the 2-dose series (1+1 vaccination schedule), with the first dose (priming dose) being given at 6-7 months of age to MenACWY- naïve healthy infants and the second dose (booster dose) given at 12-13 months of age. This study will also describe additional immunogenicity parameters and safety of MenACYW conjugate vaccine and Nimenrix® in the same population of participants.

DETAILED DESCRIPTION:
The study duration will be approximately 7 to 8.5 months (at least 7 months per participant).

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 7 months on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history, physical examination and judgment of the Investigator

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) within the past 3 months
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal infection during the study (specifically but not limited to participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease)
* Personal history of Guillain-Barré syndrome
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention(s) used in the study or to a product containing any of the same substances
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of any vaccine (including COVID-19) and Meningococcal B vaccines) in the 4 weeks preceding the first and second study intervention administration or planned receipt of any vaccine (including COVID-19 and Meningococcal B vaccines) in the 4 weeks following any study intervention administration except for influenza vaccination, which may be received at least 2 weeks before or 2 weeks after the study interventions. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal A, C, W, or Y disease with either the trial vaccine or another vaccine (i.e., mono- or quadrivalent meningococcal conjugate vaccine) containing serogroups A, C, Y, or W.

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) of Antibodies against meningococcal serogroups A, C, W and Y | 30 days after dose 2 (booster dose) (+14 days)
  Geometric mean titers after a 2-dose serie measured by serum bactericidal assays using human complement (hSBA)
Vaccine Seroresponse to meningococcal serogroups A, C, W and Y assessed by hSBA | 30 days after dose 2 (booster dose) (+14 days)
  Vaccine seroresponse after a 2-dose serie measured by hSBA

SECONDARY OUTCOMES:
hSBA antibody titers ≥ 1:8 against meningococcal serogroups A, C, W and Y | 30 days after dose 1 (priming dose) (+14 days)
  % of participants achieving antibody titers measured by hSBA ≥ predefined threshold of 1:8
hSBA antibody titers against meningococcal serogroups A, C, W and Y | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days)
  Antibody titers are measured by hSBA and summarized as geometric mean titers (GMTs)
hSBA antibody titers ≥ several pre-defined thresholds against meningococcal serogroups A, C, W and Y | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days
  Antibody titers are measured by hSBA and summarized as % of participants achieving antibody titers ≥ predefined thresholds
Percentage of Participants who achieved ≥4-fold rise in antibody titers over baseline measured by hSBA | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers 12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days
hSBA meningococcal serogroups A, C, W and Y vaccine seroresponse | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days
  Vaccine seroresponse defined as follows: For a participant with a pre-vaccination titer < 1:8, a post vaccination titer ≥ 1:16 and for a participant with a pre-vaccination titer ≥ 1:8, a post vaccination titer at least 4-fold greater than the pre vaccination titer
Rabbit complement (rSBA) antibody titers against meningococcal serogroups A, C, W, and Y | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days
rSBA antibody titers ≥ several pre-defined thresholds against meningococcal serogroups A, C, W and Y | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers 12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days
Percentage of Participants who achieved ≥4-fold rise in antibody titers over baseline measured by rSBA | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days
rSBA meningococcal serogroups A, C, W and Y vaccine seroresponse | For infants 6-7 months old: Before and 30 days after dose 1 (priming dose) (+14 days) For toddlers 12-13 months old: Before and 30 days after dose 2 (booster dose) (+14 days)
  Vaccine seroresponse defined as follows: For a participant with a pre-vaccination titer < 1:8, a post vaccination titer ≥ 1:32 and for a participant with a pre-vaccination titer ≥ 1:8, a post vaccination titer at least 4-fold greater than the pre vaccination titer
Number of participants with immediate adverse events (AEs) | Within 30 minutes after each vaccination
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions or systemic reactions | Within 7 days after each vaccination
  Pre-defined solicited injection site reactions and systemic reactions that are pre-listed in the diary cards and CRF
Number of participants with unsolicited AEs | Up to 30 days after each vaccination
  AEs other than solicited reactions
Number of participants with serious adverse events (SAEs) | From baseline to up to 7 months
  SAEs (including adverse events of special interest [AESIs]) reported throughout the study

CONTACTS AND LOCATIONS:
Locations (45):
- Czechia (3):
  - Investigational Site Number : 2030002, České Budějovice
  - Investigational Site Number: 2030001, České Budějovice
  - Investigational Site Number: 2030005, Prague
- Denmark (6):
  - Investigational Site Number: 2080007, Aalborg
  - Investigational Site Number: 2080004, Aarhus
  - Investigational Site Number: 2080006, Herlev
  - Investigational Site Number : 2080005, Hjørring
  - Investigational Site Number: 2080002, Odense
  - Investigational Site Number: 2080001, Zeeland
- Finland (8):
  - Investigational Site Number: 2460005, Espoo
  - Investigational Site Number: 2460002, Helsinki
  - Investigational Site Number: 2460011, Helsinki
  - Investigational Site Number: 2460006, Jaarvenpa
  - Investigational Site Number : 2460003, Kokkola
  - Investigational Site Number: 2460007, Oulu
  - Investigational Site Number: 2460004, Tampere
  - Investigational Site Number: 2460012, Turku
- Germany (9):
  - Investigational Site Number: 2760007, Erfurt
  - Investigational Site Number: 2760004, Herxheim
  - Investigational Site Number: 2760003, Hürth
  - Investigational Site Number: 2760001, Mönchengladbach
  - Investigational Site Number: 2760011, Mönchengladbach
  - Investigational Site Number: 2760005, Schönau am Königssee
  - Investigational Site Number: 2760008, Schweigen-Rechtenbach
  - Investigational Site Number: 2760010, Wolfsburg
  - Investigational Site Number : 2760009, Worms
- Poland (15):
  - Investigational Site Number : 6160001, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number: 6160003, Bydgoszcz
  - Investigational Site Number: 6160008, Bydgoszcz
  - Investigational Site Number: 6160017, Bydgoszcz
  - Investigational Site Number: 6160015, Krakow
  - Investigational Site Number: 6160021, Krakow
  - Investigational Site Number: 6160012, Luboń
  - Investigational Site Number: 6160011, Siemianowice Śląskie
  - Investigational Site Number: 6160007, Torun
  - Investigational Site Number: 6160014, Trzebnica
  - Investigational Site Number: 6160022, Warsaw
  - Investigational Site Number: 6160010, Wroclav
  - Investigational Site Number: 6160002, Wroclaw
  - Investigational Site Number: 6160016, Łęczna
  - Investigational Site Number: 6160004, Łomianki
- Romania (4):
  - Investigational Site Number : 6420001, Bucharest
  - Investigational Site Number : 6420003, Bucharest
  - Investigational Site Number: 6420002, Bucharest
  - Investigational Site Number: 6420005, Călăraşi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: MEQ00089 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25619&tenant=MT_SNY_9011